CLINICAL TRIAL: NCT03897803
Title: Elastography as a Follow up Imaging Tool in Patients With Idiopathic Inflammatory Myopathies
Brief Title: Elastography in Patients With Idiopathic Inflammatory Myopathies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed Ahmed Salaheldeen Hassan, Assistant professor, Benha University
Other Study IDs: BenhaU2022019
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group (I):juvenile dermatomyositis (JDM): Group (I): twenty children diagnosed to have juvenile dermatomyositis (JDM) Who will be evaluated using using strain elastography to assess muscle stiffness at baseline and after 4 months.
  .
  Interventions: Diagnostic Test: strain elastography
- Group (II):idiopathic inflammatory myopathies(IIM): Group (II): twenty adults diagnosed to have idiopathic inflammatory myopathies(IIM) Who will be evaluated using using strain elastography to assess muscle stiffness at baseline and after 4 months.
  * •
  Interventions: Diagnostic Test: strain elastography
- Group (III): juvenile control group: 20 healthy children matching age and sex as first control group to children with JDM .Who will be evaluated at baseline using using strain elastography to assess muscle stiffness .
  .
  Interventions: Diagnostic Test: strain elastography
- Group (VI):adult control group: 20 healthy adults matching age and sex as second control group to adults with IIM. Who will be evaluated at baseline using using strain elastography to assess muscle stiffness .
  Interventions: Diagnostic Test: strain elastography

INTERVENTIONS:
Diagnostic Test: strain elastography — strain elastography as apart of muscle ultrasound examination of the biceps brachii and rectus femoris muscles will be performed to the patients and control groups at baseline evaluation and after 4 months follow up in the patients groups only.

SUMMARY:
The aim of our study was to assess the performance of compression-strain US elastography in patients with idiopathic inflammatory myopathies over time and to study these findings with clinical and functional parameters as well as biochemical and electromyographic tests.

DETAILED DESCRIPTION:
This study will be carried out on four groups:

Group (I): twenty children diagnosed to have idiopathic inflammatory myopathies(IIM)

* Group (II): twenty adults diagnosed to have IIM
* Group (III):20 healthy children matching age and sex as first control group to children with IIM .
* Group (VI):20 healthy adults matching age and sex as second control group to adults with IIM.

All patients will be evaluated at baseline at & 4-months follow up using Semi-Quantitative strain elastography

ELIGIBILITY:
Inclusion Criteria:

* to fulfill criteria of diagnosis of childhood and adult idiopathic inflammatory myopathies

Exclusion Criteria:

* Patients with age less than 2 years were excluded from the study due to inability to perform manual muscle testing and functional scales.
* The presence of a associated illness that may result in nerve or muscle affection

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be carried out on four groups:
  Group (I): thirty children diagnosed to have idiopathic inflammatory myopathies(IIM)
  * Group (II): thirty adults diagnosed to have IIM
  * Group (III):30 healthy children matching age and sex as first control group to children with IIM .
  * Group (VI):30 healthy adults matching age and sex as second control group to adults with IIM.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Manual muscle testing | 6 months
  Kendall's 0 -10 point scale measures strength of each muscle group score 0 is the weakest (worst) and 10 is the strongest (best). The following muscles were tested bilaterally: the biceps brachii muscle (BB), the forearm flexors(FF), the rectus femoris muscle (RF), the tibialis anterior muscle (TA)
Serum creatine kinase (CK) levels | 6 months
  CK measured in U/L using ELISA
Serum Lactate dehydrogenase (LDH) levels | 6 months
  LDHmeasured in IU/L using ELISA
alanine aminotransferase (ALT) | 6 months
  ALT measured in U/L using ELISA
Aspartate aminotransferase (AST) | 6 months
  AST measured in U/L using ELISA
motor unit potential (MUP) duration | 6 months
  quantitative electromyography (QEMG) in the most affected rectus femoris and biceps brachii muscles will be performed and The motor unit potentials will be reviewed offline for the needle-detected EMG signals will be analyzed by the device software for the MUP duration measured in milliseconds.
motor unit peak-to-peak amplitude | 6 months
  quantitative electromyography (QEMG) in the most affected rectus femoris and biceps brachii muscles will be performed and The motor unit potentials will be reviewed offline for the needle-detected EMG signals will be analyzed by the device software for the peak-to-peak amplitude measured in microvolt
motor unit area to amplitude ratio (AAR) | 6 months
  quantitative electromyography (QEMG) in the most affected rectus femoris and biceps brachii muscles will be performed and The motor unit potentials will be reviewed offline for the needle-detected EMG signals will be analyzed by the device software for the motor unit AAR .
muscle echo intenisity (EI) | 6 MONTHS
  EI is assessed during muscle ultrasound evaluation means of computer-assisted grayscale histogram analysis of Adobe Photoshop . echo intensity was calculated based on a histogram analysis which expresses every pixel as a value between 0 (black) and 255 (white)..he following muscles were tested bilaterally: the biceps brachii muscle (BB), the forearm flexors(FF), the rectus femoris muscle (RF), the tibialis anterior muscle (TA)
Childhood myositis assessment scale | 6 months
  used to assess the severity of muscle involvement in children with dermatomyositis. The scores for the 14 items are summated to give a total score ranging from 0 (worst) to 52 (best)
MYOSITIS DISEASE ACTIVITY ASSESSMENT TOOL (MDAAT) | 6 months
  The MDAAT is a combined tool that includes the Myositis Disease Activity Assessment visual analog scale (VAS) (MYOACT) and the Myositis Intention to Treat Activities Index (MITAX).it Assesses 6 extramuscular organs to produce a global extramuscular score, and the muscle score, which gives a total disease activity index score. Scores range from 0-60 for the extramuscular MYOACT score and 0-70 for the total MYOACT score, and they range from 0-54 for the Extramuscular MITAX score and 0-63 for the total MITAX score. higher scores indicates worse outcome
CHILDHOOD HEALTH ASSESSMENT QUESTIONNAIRE (CHAQ) | 6 months
  There are 30 items in the Disability Index; one item each in the Discomfort Index and Health Status Index. Score range. The range is 0-3. Higher scores reflect greater disability.
HEALTH ASSESSMENT QUESTIONNAIRE (HAQ) | 6months
  20 questions grouped into eight subscales (dressing and grooming, arising, eating, walking, hygiene, reach, grip, activities). (score = 0 to 3 with higher score means worse outcome ). The highest score for any question determines the score for the subscale in question. The HAQ disability index is calculated as the sum of the scores for various subscales,divided by the number of subscales responded to, and results in a score between 0 and 3. higher score means worse outcome
MYOSITIS DAMAGE INDEX (MDI) | 6months
  The MDI measures specific manifestations in 11 organ systems The MDI also includes a series of visual analog scales (VAS) to quantify damage severity in a given organ system. The VAS are summed together for a potential score of 0-110 with higher scores has worse prognosis
PHYSICIAN GLOBAL ACTIVITY assessment | 6 months
  visual analogue scale rating, a score of 0-10 (down to 1 decimal place) is used, higher score means worse outcome
PATIENT/PARENT GLOBAL ACTIVITY assessment | 6 months
  visual analogue scale rating, a score of 0-10 (down to 1 decimal place) is used, higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Waleed A Hassan, MD, Principal Investigator — Benha university- Qaluibya- Egypt
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt